CLINICAL TRIAL: NCT00003339
Title: A Randomized Phase II Trial of a Vaccine Combining Tyrosinase/gp100 Peptides Emulsified With Montanide ISA 51 With and Without Interleukin-12 for Patients With Resected Stages III and IV Melanoma
Brief Title: Vaccine Therapy With or Without Interleukin-12 in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066310 (10M-97-3); LAC-USC-10M973; NCI-G98-1432; NCI-T97-0099
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: recurrent intraocular melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — incomplete Freund's adjuvant; Interleukin-12 Subunit p35

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: recombinant interleukin-12
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines made from a person's cancer cells may make the body build an immune response that will kill tumor cells. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating white blood cells to kill melanoma cells.

PURPOSE: Randomized phase II trial to determine the effectiveness of vaccine therapy given with interleukin-12 in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate immune reactivity to tyrosinase and gp100 peptides emulsified with Montanide ISA-51 (ISA-51) with or without interleukin-12 following surgical resection in HLA-A2 positive patients with stage III or IV melanoma.

OUTLINE: This is a randomized, parallel study. Patients are stratified by prior therapy (immunotherapy or chemotherapy vs surgery only). Patients are randomized to receive 1 of 2 treatment arms: Arm I: Following surgery, patients receive tyrosinase and gp100 peptides emulsified with Montanide ISA-51 (ISA-51) subcutaneously (SQ) once weekly during weeks 0, 2, 4, 6, 10, 14, 18, and 26 for a total of 8 vaccinations. Arm II: Following surgery, patients receive treatment as in Arm I followed by interleukin-12 SQ once weekly during weeks 0, 2, 4, 6, 10, 14, 18, and 26 for a total of 8 vaccinations. Patients are followed at 2-4 weeks, then every 3 months for 2 years after resection, then every 6 months for 3 years, and then yearly if without evidence of disease.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage III or IV cutaneous or ocular melanoma that can be completely resected or rendered free of disease but is at high risk of recurrence OR Recurrent disease following interferon alfa or ineligible for or refused interferon alfa HLA-A2 positive Tumor tissue must be available for analysis of gp100/tyrosinase expression Detectable expression of one or the other antigen not required

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Absolute granulocyte count at least 1,500/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: No major cardiovascular illness Pulmonary: No major respiratory illness (e.g., pneumonia) Gastrointestinal: No major gastrointestinal illness Other: Not pregnant or nursing No major systemic infection (e.g., sepsis) No coagulation or bleeding disorder HIV negative Hepatitis B surface antigen negative Hepatitis C surface antigen negative No history of uveitis or autoimmune inflammatory eye disease No active autoimmune disease Not allergic to Montanide ISA-51 No active second malignancy within the past 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 1 month since prior biologic therapy Chemotherapy: At least 1 month since prior chemotherapy, including adjuvant therapy Endocrine therapy: At least 1 month since prior endocrine therapy No concurrent steroid therapy Radiotherapy: At least 1 month since prior radiotherapy Surgery: See Disease Characteristics At least 1 month since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1998-11; Primary Completion 1999-11 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (2):
- United States (2):
  - Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California